CLINICAL TRIAL: NCT03736759
Title: Resistance Exercise to Improve Vaccine Outcomes in Older Adults
Brief Title: Resistance Exercise to Improve Flu Vaccine for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Emily C Lavoy, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00000542; R03AG052778 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Influenza, Human
Keywords: exercise; vaccine; older adults
MeSH Terms: conditions — Influenza, Human; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise and vaccine in same arm (Experimental): 20 min eccentric resistance exercise of deltoid and biceps brachii in non-dominant arm, followed immediately by intramuscular injection of seasonal quadrivalent influenza vaccine in non-dominant arm
  Interventions: Behavioral: Exercise
- Exercise and vaccine in different arms (Active Comparator): 20 min eccentric resistance exercise of deltoid and biceps brachii in dominant arm, followed immediately by intramuscular injection of seasonal quadrivalent influenza vaccine in non-dominant arm
  Interventions: Behavioral: Exercise
- vaccine only (No Intervention): 20 min rest followed immediately by intramuscular injection of seasonal quadrivalent influenza vaccine in non-dominant arm

INTERVENTIONS:
Behavioral: Exercise — 10 sets of 5 repetitions of 80% of calculated one-repetition maximum weight of lateral side arm raise and biceps curls, alternating
  Arms: Exercise and vaccine in different arms; Exercise and vaccine in same arm

SUMMARY:
This study evaluates whether resistance exercise will improve immune responses to the seasonal influenza vaccine in older adults. One third of the participants will perform exercise in the arm that receives the vaccine, one third of the participants will perform the same exercise in the arm that does not receive the vaccine, and one third will only receive the vaccine.

DETAILED DESCRIPTION:
Resistance exercise, particularly novel eccentric exercise, recruits immune cells to the targeted muscle. The exercises selected here targets the deltoid and biceps brachii muscles-those same muscles that the flu vaccine is delivered to during typical vaccination.

ELIGIBILITY:
Inclusion Criteria:

* non-frail older adult (≥65 years old) of any sex and race/ethnicity
* non-smokers (>10 yrs)
* meets American College of Sports Medicine criteria for participation in exercise
* US resident

Exclusion Criteria:

* underlying medical problems that contraindicate supervised resistance exercise
* past or present history of autoimmune disease, HIV, hepatitis, stroke, or cardiovascular disease
* current debilitating arthritis of the shoulder
* central or peripheral nervous disorders
* bedridden in the past three months
* history of vaccine-related allergies, or severe egg allergy;
* physician-confirmed influenza infection in the prior year
* regular user of corticosteroids
* functional or cognitive impairment that would limit exercise performance or prohibit informed consent
* blood pressure greater than 160/90
* participation in resistance arm exercises in the prior 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Cell mediated immunity change at 6 weeks post-vaccine | baseline and 6 weeks
  The change in the peripheral blood mononuclear cell response to overnight ex vivo culture with the seasonal quadrivalent vaccine detected via Interferon-gamma ELISPOT will be calculated from baseline at 6 weeks post-vaccine
Antibody titer change at 6 weeks post-vaccine | baseline and 6 weeks
  The change in influenza-specific antibody titers in serum measured by hemagglutination inhibition assay will be calculated from baseline at 6 weeks post-vaccine
Cell mediated immunity change at 6 months post-vaccine | baseline and 6 months
  The change in the peripheral blood mononuclear cell response to overnight ex vivo culture with the seasonal quadrivalent vaccine detected via Interferon-gamma ELISPOT will be calculated from baseline at 6 months post-vaccine
Antibody titer change at 6 months post-vaccine | baseline and 6 months
  The change in influenza-specific antibody titers in serum measured by hemagglutination inhibition assay will be calculated from baseline at 6 months post-vaccine

SECONDARY OUTCOMES:
Muscle soreness | 7 days
  Self-reported pain in upper arm shoulder/ region of both arms collected once daily for 7 days after vaccination. Item will be scored 0-10 (0= no pain; 10= worst possible pain).
Influenza-like symptoms | Measured monthly for six months
  Self-report symptoms of influenza infection, guided by an influenza self-screening questionnaire( modified from University of California Davis Student Health and Counseling Service influenza self-screening questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Emily C LaVoy, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Elzayat MT, Markofski MM, Simpson RJ, Laughlin M, LaVoy EC. No Effect of Acute Eccentric Resistance Exercise on Immune Responses to Influenza Vaccination in Older Adults: A Randomized Control Trial. Front Physiol. 2021 Aug 12;12:713183. doi: 10.3389/fphys.2021.713183. eCollection 2021. PMID 34456752